CLINICAL TRIAL: NCT04484077
Title: A PHASE I STUDY OF hCT-MSC, AN UMBILICAL CORD-DERIVED MESENCHYMAL STROMAL CELL PRODUCT, IN ADULTS WITH AUTISM SPECTRUM DISORDER
Brief Title: hCT-MSC Infusion in Adults With Autism Spectrum Disorder
Acronym: AIMs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Collaborators: The Marcus Foundation (Other)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Jerome Harris Distinguished Professor of Pediatrics; Professor of Pathology; Director, Marcus Center for Cellular Cures; Director, Pediatric Blood and Marrow Transplant Program; Director, Carolinas Cord Blood Bank, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00104691
Record Dates: First submitted 2020-07-16; First posted 2020-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: autism; MSC; hCT-MSC; mesenchymal stromal cells
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- hCT-MSC infusion (Experimental): A single, intravenous infusion of hCT-MSCs. Targeted dose is 2x10^6 cells/kg with a maximum dose of 10 x 10^7 cells/kg.
  Interventions: Biological: hCT-MSC

INTERVENTIONS:
Biological: hCT-MSC — 2x10^6 hCT-MSC/kg suspended in plasmalyte-A, 5% HSA, and residual DMSO/dextran administered intravenously over 30-60 minutes via syringe pump

SUMMARY:
The purpose of the study is to determine the safety and tolerability of a single intravenous dose of Human Umbilical Cord Tissue Derived Mesenchymal Stromal Cells (hCT-MSC) in adults with autism spectrum disorder (ASD). hCT-MSC is a cell product isolated from umbilical cord tissue. The cells from the cord tissue are processed and expanded in the laboratory and then infused intravenously in a single dose per participant. Participants will be ages 18-35 years, with ASD and a full-scale IQ >70 without an identified genetic cause of autism. Participants will have an in-person baseline visit and remote follow up visits at 6 and 12 months. In addition to the primary endpoints evaluating safety, the study will evaluate changes in social communications skills after hCT-MSC administration.

DETAILED DESCRIPTION:
This is a prospective, open label, phase one study to determine the safety and tolerability of a single intravenous dose of Human Umbilical Cord Tissue Derived Mesenchymal Stromal Cells (hCT-MSC) in adults with autism spectrum disorder (ASD). hCT-MSCs are manufactured from umbilical cord tissue donated by healthy mothers delivering full term babies via Cesarean Section. The cells are extracted from the cord tissue, expanded and cryopreserved (frozen). One dose of 2x10^6 cells/kg (maximum of 10 x 10^7) will be administered intravenously to each participant in this study.

It is hypothesized that immune dysregulation and/or abnormal neuronal connectivity that adversely affects normal brain development may cause core symptomatology observed in individuals with ASD. Mesenchymal stromal cells (MSC) have demonstrated a multitude of immunomodulatory effects which are thought to be carried out via paracrine and trophic signaling. While MSCs modulate the immune response, MSCs themselves have low immunogenicity (the body does not have a strong immune reaction against them) and they do not permanently engraft in the recipient.

Adults ages 18 to less than 35 years with ASD will be eligible to participate. All participants will have a screening visit that includes clinical evaluations to verify cognitive abilities and confirmation of eligibility.

One dose of 2x10^6 cells/kg (maximum of 10 x 10^7) will be administered intravenously to each participant at a baseline visit. Participants will be admitted to the infusion center on the day of their baseline visit and vital signs (heart rate, blood pressure, temperature, respiratory rate) will be measured. Participants may request anti-anxiety medication prior to IV placement if desired. A peripheral IV will be placed and prior to the infusion, premedications (Benadryl, Solumedrol, 0.5mg/kg each) will be administered. The hCT-MSCs product will be administered intravenously over 30-60 minutes. Pulse oximetry will be monitored continuously throughout the infusion and IV fluid maintenance will be given. Participants will be discharged after 1 hour, providing all vital signs are at their baseline and they are asymptomatic with no evidence of toxicity. Participants will be evaluated the day after the infusion to assess for any infusion-related adverse reactions or complications. A phone call or email will be done to assess safety of the infusion 7-10 days after the infusion. Remote follow up will be conducted 6 months and one year after infusion. The Medical and Behavioral History Questionnaire assessing adverse events will be obtained at baseline, 6 and 12-months.

The main endpoint is safety, and acute infusion reactions, incidence of infections, and markers of alloimmunization will be assessed. Social communication will be assessed at baseline and 6 months post product administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 to < 35 years (34 years, 364 days) at the time of consent
2. Confirmed pre-existing diagnosis of ASD in the individual's educational and/or medical record
3. Fragile X testing performed and negative; CMA and/or whole exome sequencing performed and results not linked to autism diagnosis
4. Stable on current psychiatric medication regimen (dose and dosing schedule) for at least 2 months prior to infusion of study product, with no intention of changing or beginning new psychiatric medications or behavioral treatments during the duration of the study.
5. Normal absolute lymphocyte count (≥1200/uL for African American participants and ≥1500/uL for all other participants)
6. General Ability Index of ≥70, confirmed through cognitive testing completed by study personnel to establish eligibility
7. Participant and Parent are English speaking
8. Able to travel to Duke University for baseline visit.
9. Participant has a parent who spends four or more hours a week with the participant, who is able and willing to participate in study visits and interim surveys and interviews
10. Informed consent of the participant and parent (participants must have legal authority regarding their own medical care and a parent or legally authorized representative may not consent on their behalf)

Exclusion Criteria

1. General:

   1. Review of medical records indicates ASD diagnosis and IQ > 70 unlikely.
   2. Known or suspected diagnosis of any of the following coexisting psychiatric conditions: bipolar disorder, schizophrenia, Tourette syndrome, and/or any co-occurring psychiatric disorder that the investigator believes would interfere with accurate completion of study instruments and/or current (within the past year) evidence of suicidality as assessed by an interview with participant and/or parent which includes the Columbia Suicide Severity Rating Scale, and a review of responses on the Behavioral and Symptom Identification Scale (BASIS-24).
   3. Screening data or in-person evaluations suggest that participant would not be able to comply with the requirements of the study procedures as assessed by the study team
   4. Parent and/or participant is unwilling or unable to commit to participation in all study-related assessments, including protocol follow up
   5. Sibling is enrolled in this (Duke AIMs) study
2. Genetic:

   1. Records indicate that the participant has a known genetic syndrome such as (but not limited to) Fragile X syndrome, neurofibromatosis, Rett syndrome, tuberous sclerosis, PTEN mutation, cystic fibrosis, muscular dystrophy or a genetic defect definitively known to be associated with ASD
   2. Known pathogenic mutation or copy number variation (CNV) associated with ASD (e.g., 16p11.2, 15q13.2, 2q13.3)
3. Infectious:

   1. Known active CNS infection
   2. Evidence of uncontrolled infection based on records or clinical assessment
   3. Known HIV positivity
   4. Exposure to COVID-19 in the preceding 14 days or positive COVID-19 test in the previous 28 days. Subjects with a past history of infection with COVID-19 must be symptom-free for 14 days prior to the initial visit.
4. Medical:

   1. Known metabolic disorder
   2. Known mitochondrial dysfunction
   3. History of unstable epilepsy or uncontrolled seizure disorder, infantile spasms, Lennox Gastaut syndrome, Dravet syndrome, or other similar chronic seizure disorder
   4. Active malignancy or prior malignancy that was treated with chemotherapy
   5. History of a primary immunodeficiency disorder
   6. History of autoimmune cytopenias (i.e., ITP, AIHA)
   7. Coexisting medical condition that would place the participant at increased risk for complications of study procedures
   8. Concurrent genetic or acquired disease or comorbidity(ies) that could require a future stem cell transplant
   9. Significant sensory (e.g., blindness, deafness, uncorrected hearing impairment) or motor (e.g., cerebral palsy) impairment
   10. Impaired renal or liver function as determined by serum creatinine >1.5mg/dL or total bilirubin >1.3mg/dL, except in participants with known Gilbert's disease
   11. Significant hematologic abnormalities defined as: Hemoglobin <10.0 g/dL, Platelets <150 x 10e9/uL, WBC <3,000 cells/mL, ALC <1200/uL for African Americans or <1500/uL for all other participants.
   12. Evidence of clinically relevant physical dysmorphology indicative of a genetic syndrome as assessed by the PIs or other investigators, including a medical geneticist and psychiatrists trained in identifying dysmorphic features associated with neurodevelopmental conditions.
   13. Current pregnancy and unwillingness to use adequate birth control for 3 months after the final study product infusion.
5. Current/Prior Therapy:

   a. Availability of a banked, qualified autologous cord blood unit or parent deferred use of qualified, autologous cord blood unit b. History of prior cell therapy c. Current or prior use of IVIG or other anti-inflammatory medications with the exception of NSAIDs d. Current or prior immunosuppressive therapy i. No systemic steroid therapy that has lasted >5 days within 4 weeks, prior to enrollment. Topical and inhaled steroids are permitted.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Incidence of infusion reactions | Baseline through 10 days post infusion
  cumulative incidence as measured by clinical examination and patient interview
Incidence of product-related infections | Baseline through 12 months
  cumulative incidence as measured by patient interview and questionnaire
Evidence of formation of anti-HLA antibodies | Baseline, 6 months, 12 months
  change from baseline to 6 and 12 months post infusion as measured by PRA testing
Incidence of graft vs. host disease | Baseline through 12 months
  cumulative incidence as measured by patient interview and questionnaire
Incidence of unexpected adverse events, by severity and relation to study | Baseline through 12 months
  cumulative incidence as measured by patient questionnaire and clinical labs

SECONDARY OUTCOMES:
The Vineland Adaptive Behavior Scale Interview, 3rd Edition, Comprehensive interview form | Baseline and 6 months
  Change from baseline to six months in the Combined Socialization Standard Score based on parent report. Scores range from 20 to 140. Higher scores indicate a higher functioning level

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Sun, MD, Principal Investigator — Duke University; Joanne Kurtzberg, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No